CLINICAL TRIAL: NCT00003571
Title: Tumor Replication Error (RER) Status and Outcome in a Colon Cancer Adjuvant Chemotherapy Trial
Brief Title: Gene Testing in Patients With Colon Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9865; U10CA031946 (NIH); CLB-9865; CDR0000066637 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-07-15 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; adenocarcinoma of the colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of tumor and normal tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Samples of tumor and normal tissue: Samples of tumor and normal tissue are obtained from CALGB 8896 patients. The samples are tested for somatic mutations and tumor replication error (RER) tumor status. Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.
  Interventions: Genetic: mutation analysis; Genetic: tumor replication error analysis

INTERVENTIONS:
Genetic: mutation analysis
Genetic: tumor replication error analysis

SUMMARY:
RATIONALE: Analyzing the structure of genes found in a person's cancer cells may help doctors improve methods of treating patients with colon cancer.

PURPOSE: Clinical trial to study the genes of patients treated with chemotherapy for colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the relationship between disease free survival, overall survival, and tumor replication error status for patients who have received adjuvant chemotherapy for colon cancer on CALGB protocol 8896.
* Determine the prognostic and predictive values for response to this therapy in these patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients who received chemotherapy for colon cancer as part of CALGB protocol 8896
* Underwent an initial resection for adenocarcinoma of the colon and were determined to have a high risk of tumor recurrence based upon nodal disease or local extension of tumor with obstruction or perforation due to tumor
* Surgical specimen blocks available, including tumor tissue and normal tissue

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously enrolled on CALGB-8896.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 1998-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
disease free survival | Up to 10 years

SECONDARY OUTCOMES:
overall survival | Up to 10 years
tumor replication error status | Up to 10 years
determine the prognostic and predictive values for response to this therapy | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Monica M. Bertagnolli, MD, Study Chair — Dana-Farber/Brigham and Women's Cancer Center
Locations (44):
- United States (44):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Background] Goel A, Arnold CN, Niedzwiecki D, Carethers JM, Dowell JM, Wasserman L, Compton C, Mayer RJ, Bertagnolli MM, Boland CR. Frequent inactivation of PTEN by promoter hypermethylation in microsatellite instability-high sporadic colorectal cancers. Cancer Res. 2004 May 1;64(9):3014-21. doi: 10.1158/0008-5472.can-2401-2. PMID 15126336
- [Background] Goel A, Arnold CN, Niedzwiecki D, Chang DK, Ricciardiello L, Carethers JM, Dowell JM, Wasserman L, Compton C, Mayer RJ, Bertagnolli MM, Boland CR. Characterization of sporadic colon cancer by patterns of genomic instability. Cancer Res. 2003 Apr 1;63(7):1608-14. PMID 12670912
- [Result] Arnold CN, Goel A, Compton C, Marcus V, Niedzwiecki D, Dowell JM, Wasserman L, Inoue T, Mayer RJ, Bertagnolli MM, Boland CR. Evaluation of microsatellite instability, hMLH1 expression and hMLH1 promoter hypermethylation in defining the MSI phenotype of colorectal cancer. Cancer Biol Ther. 2004 Jan;3(1):73-8. doi: 10.4161/cbt.3.1.590. Epub 2004 Jan 5. PMID 14726676
- [Result] Goel A, Arnold CN, Tassone P, Chang DK, Niedzwiecki D, Dowell JM, Wasserman L, Compton C, Mayer RJ, Bertagnolli MM, Boland CR. Epigenetic inactivation of RUNX3 in microsatellite unstable sporadic colon cancers. Int J Cancer. 2004 Dec 10;112(5):754-9. doi: 10.1002/ijc.20472. PMID 15386381